CLINICAL TRIAL: NCT05817526
Title: Assessment of Collagen Loaded With Bone Marrow Aspirate Concentrate Versus Autograft on Marginal Bone Changes Around Immediate Implants in Esthetic Zone. A Randomized Controlled Clinical Trial
Brief Title: BMAC Loaded Collagen Jumping the Gap Around Immediate Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, Lecturer of oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMAC around immediate implants
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Implant Site Reaction; Dental Implantation
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMAC/ collagen (Active Comparator): Bone marrow aspirate concentrate loaded on collagen utilization for filling peri-implant gap around immediate dental implants in the Maxillary esthetic zone
  Interventions: Drug: BMAC/ collagen
- Autograft (Active Comparator): Autograft harvested from chin utilization for filling peri-implant gap around immediate dental implants in the Maxillary esthetic zone
  Interventions: Procedure: Autograft harvesting from chin

INTERVENTIONS:
Drug: BMAC/ collagen — Bone marrow aspirate concentrate loaded on collagen in the peri-implant defect
  Other Names: Bone marrow aspirate concentrate group
  Arms: BMAC/ collagen
Procedure: Autograft harvesting from chin — Autograft
  Other Names: Autograft group
  Arms: Autograft

SUMMARY:
The present study aims to evaluate the effect of utilization of BMAC/ collagen on marginal bone changes around immediate implants in the esthetic zone of maxilla.

Methodology: Twenty dental implants will be installed in the esthetic zone and patients will be randomly divided into two groups:

study group: The jumping gap surrounding the immediate implants will be grafted with BMAC/collagen, whereas in the control group, autograft from the chin will be used to fill the defect. Cone beam CT (CBCT) will be requested Preoperative, immediate and 4 months Postoperative for assessment of marginal bone changes around implants.

.

DETAILED DESCRIPTION:
The aim of present study is to evaluate the effect of utilization of bone marrow aspirate concentrate (BMAC) loaded on collagen on the marginal bone changes around immediate implants in the esthetic zone of maxilla.

Methodology: Twenty dental implants will be installed in patients suffering from non- restorable teeth in esthetic zone.

Patients will be randomly divided into two equal groups:

study group: The jumping gap surrounding the immediate implants will be grafted with bone marrow aspirate concentrate loaded on collagen, whereas in the control group, autogenous bone graft from the chin will be used to fill the peri-implant defect. CBCT will be requested Preoperative, immediate and 4 months Postoperative for assessment of marginal bone changes around dental implants.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non- restorable teeth in esthetic zone
* Patients above 18 us
* Highly motivated patients.

Exclusion Criteria:

* patients with systemic diseases • immunocompromised patients . Patients with bleeding disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Marginal bone changes | 4 months
  Buccal bone height

CONTACTS AND LOCATIONS:
Overall Officials: Eman Said, Study Director — Lecturer at Faculty of Dentistry, Cairo University
Locations (1):
- Walaa Kadry, Cairo, Egypt